CLINICAL TRIAL: NCT02290717
Title: Fractional Laser Abrasion in Combination With UVB Therapy in Vitiligo Patients: a Randomized Controlled Study.
Brief Title: Fractional Laser in Combination With UVB Therapy in Vitiligo Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty including patients
Sponsor: Netherlands Institute for Pigment Disorders (Other)
Responsible Party: Principal Investigator, JELommerts, MSc MD, Netherlands Institute for Pigment Disorders
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL45970.018.13
Record Dates: First submitted 2014-11-07; First posted 2014-11-14 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Vitiligo
Keywords: ultraviolet therapy; non segmental; vitiligo; topical corticosteroid; laser; fractional; CO2; carbon dioxide; UVB
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Laser+fluticason+UVB (Experimental): The treatment site will be superficially abraded using an ablative fractional laser (10,600nm CO2 laser). 5 days after laser therapy topical steroids (fluticasone cream) 4 times a week will be applied on the treatment site until the end of the study.
  Interventions: Device: Fractional CO2 laser; Other: NB-UVB therapy; Drug: Fluticasone Propionate Cream 0.05%
- Laser+UVB (Experimental): In one session the treatment site will be superficially abraded using an ablative fractional laser (10,600nm CO2 laser).
  Interventions: Device: Fractional CO2 laser; Other: NB-UVB therapy
- UVB (Active Comparator): As control site, 1 similar depigmented lesion will be used. This site will receive the same NB-UVB treatment as sites 1 and 2.
  Interventions: Other: NB-UVB therapy

INTERVENTIONS:
Device: Fractional CO2 laser
  Arms: Laser+UVB; Laser+fluticason+UVB
Other: NB-UVB therapy — NB-UVB therapy (according to the standard treatment protocol of the SNIP, which the patient is already been treated with) will be continued for both treated and control sites during 6 months.
Drug: Fluticasone Propionate Cream 0.05% — 4 times a week (standard IPD protocol)
  Arms: Laser+fluticason+UVB

SUMMARY:
Rationale: Vitiligo is a common skin disorder that can impair a patient's quality of life. Many depigmented lesions in vitiligo patients remain therapy resistant for medical treatment. Therefore new therapeutic options in these patients are necessary. Currently, dermabrasion by conventional or fractional laser therapy in combination with NB-UVB therapy and steroids appears to be effective in therapy resistant areas. However, little literature on this combination is available.

Objectives: To assess the efficacy and patient safety of (1)fractional CO2-laser treatment in combination with NB- UVB,(2) fractional CO2-laser treatment in combination with NB- UVB and topical corticosteroids versus NB-UVB treatment alone(3) Study design: Prospective observer blinded randomised intra-patient controlled study.

Study population: 23 patients ≥ 18 years with non segmental vitiligo who receive NB-UVB treatment at the Netherlands Institute for Pigment Disorders (SNIP) at the Academic Medical Centre University of Amsterdam. We will include patients with 3 depigmented lesions that are resistant to NB- UVB treatment after 3 to 6 months.

Methods: Three NB-UVB resistant depigmented regions on the trunk or extremities will be randomly allocated to;(1) NB-UVB treatment in combination with fractional CO2 laser abrasion, or (2) NB-UVB treatment in combination with fractional CO2 laser abrasion and topical steroids, or (3) NB-UVB treatment alone. NB-UVB treatment and topical steroids will be given according to the standard treatment protocol of the SNIP and continued for at least 6 months. Two and 6 months after the laser treatment, the percentage of repigmentation of the lesions will be assessed.

ELIGIBILITY:
Inclusion criteria

* Patients with non segmental (generalised) vitiligo visiting the Netherlands Institute for Pigment Disorders
* receiving NB- UVB treatment for 3 to 6 months
* Age >18 years
* At least 3 therapy resistant vitiligo lesions on the extremities or trunk larger than 5x5 cm or one vitiligo lesion on the extremities or trunk of at least 5x15 cm.
* Patient is willing and able to give written informed consent

Exclusion criteria

* Skin type I
* Recurrent HSV skin infections
* Hypertrophic scars
* Keloid
* Cardial insufficiency
* Patients who are pregnant or breast-feeding
* Patients not competent to understand what the procedures involved
* Patients with a personal history of melanoma or non-melanoma skin cancer
* Patients with atypical nevi.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Repigmentation % with sheets | 6 mo after treatment
  % of repigmentation

SECONDARY OUTCOMES:
Global assessment physician | 6 months after treatment
Global assessment patient | 6 months after treatment
Visual assessment of hyperpigmentation/hypopigmentation/scar formation | 6 months after treatment
Global assessment of repigmentation physician | 6months after treatment

OTHER OUTCOMES:
Adverse events | 6 months after treatment
Color difference between erythema and (re)pigmentation | 6 months after treatment
  with a Derma-spectrometer the difference between erythema and (re)pigmentation will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Centre, Amsterdam, Netherlands

REFERENCES:
- [Background] Garg T, Chander R, Jain A. Combination of microdermabrasion and 5-fluorouracil to induce repigmentation in vitiligo: an observational study. Dermatol Surg. 2011 Dec;37(12):1763-6. doi: 10.1111/j.1524-4725.2011.02127.x. Epub 2011 Aug 11. PMID 21834930
- [Background] Shin J, Lee JS, Hann SK, Oh SH. Combination treatment by 10 600 nm ablative fractional carbon dioxide laser and narrowband ultraviolet B in refractory nonsegmental vitiligo: a prospective, randomized half-body comparative study. Br J Dermatol. 2012 Mar;166(3):658-61. doi: 10.1111/j.1365-2133.2011.10723.x. Epub 2012 Jan 19. PMID 22050270
- [Background] Bayoumi W, Fontas E, Sillard L, Le Duff F, Ortonne JP, Bahadoran P, Lacour JP, Passeron T. Effect of a preceding laser dermabrasion on the outcome of combined therapy with narrowband ultraviolet B and potent topical steroids for treating nonsegmental vitiligo in resistant localizations. Br J Dermatol. 2012 Jan;166(1):208-11. doi: 10.1111/j.1365-2133.2011.10564.x. Epub 2011 Nov 17. PMID 21824124
- [Background] Linthorst Homan MW, Spuls PI, de Korte J, Bos JD, Sprangers MA, van der Veen JP. The burden of vitiligo: patient characteristics associated with quality of life. J Am Acad Dermatol. 2009 Sep;61(3):411-20. doi: 10.1016/j.jaad.2009.03.022. Epub 2009 Jul 3. PMID 19577331
- [Background] Ongenae K, Van Geel N, De Schepper S, Naeyaert JM. Effect of vitiligo on self-reported health-related quality of life. Br J Dermatol. 2005 Jun;152(6):1165-72. doi: 10.1111/j.1365-2133.2005.06456.x. PMID 15948977
- [Background] Alikhan A, Felsten LM, Daly M, Petronic-Rosic V. Vitiligo: a comprehensive overview Part I. Introduction, epidemiology, quality of life, diagnosis, differential diagnosis, associations, histopathology, etiology, and work-up. J Am Acad Dermatol. 2011 Sep;65(3):473-491. doi: 10.1016/j.jaad.2010.11.061. PMID 21839315
- [Background] Drake LA, Dinehart SM, Farmer ER, Goltz RW, Graham GF, Hordinsky MK, Lewis CW, Pariser DM, Skouge JW, Turner ML, Webster SB, Whitaker DC, Lowery BJ, Nordlund JJ, Grimes PE, Halder RM, Minus HR. Guidelines of care for vitiligo. American Academy of Dermatology. J Am Acad Dermatol. 1996 Oct;35(4):620-6. doi: 10.1016/s0190-9622(96)90691-x. No abstract available. PMID 8859294
- [Background] Njoo MD, Westerhof W. Vitiligo. Pathogenesis and treatment. Am J Clin Dermatol. 2001;2(3):167-81. doi: 10.2165/00128071-200102030-00006. PMID 11705094
- [Background] Taieb A, Picardo M. Clinical practice. Vitiligo. N Engl J Med. 2009 Jan 8;360(2):160-9. doi: 10.1056/NEJMcp0804388. No abstract available. PMID 19129529
- [Background] Taieb A, Alomar A, Bohm M, Dell'anna ML, De Pase A, Eleftheriadou V, Ezzedine K, Gauthier Y, Gawkrodger DJ, Jouary T, Leone G, Moretti S, Nieuweboer-Krobotova L, Olsson MJ, Parsad D, Passeron T, Tanew A, van der Veen W, van Geel N, Whitton M, Wolkerstorfer A, Picardo M; Vitiligo European Task Force (VETF); European Academy of Dermatology and Venereology (EADV); Union Europe enne des Me decins Spe cialistes (UEMS). Guidelines for the management of vitiligo: the European Dermatology Forum consensus. Br J Dermatol. 2013 Jan;168(1):5-19. doi: 10.1111/j.1365-2133.2012.11197.x. Epub 2012 Nov 2. PMID 22860621
- [Background] Lotti T, Buggiani G, Troiano M, Assad GB, Delescluse J, De Giorgi V, Hercogova J. Targeted and combination treatments for vitiligo. Comparative evaluation of different current modalities in 458 subjects. Dermatol Ther. 2008 Jul;21 Suppl 1:S20-6. doi: 10.1111/j.1529-8019.2008.00198.x. PMID 18727812
- [Background] Farajzadeh S, Daraei Z, Esfandiarpour I, Hosseini SH. The efficacy of pimecrolimus 1% cream combined with microdermabrasion in the treatment of nonsegmental childhood vitiligo: a randomized placebo-controlled study. Pediatr Dermatol. 2009 May-Jun;26(3):286-91. doi: 10.1111/j.1525-1470.2009.00926.x. PMID 19706089
- [Background] van Geel N, Ongenae K, Naeyaert JM. Surgical techniques for vitiligo: a review. Dermatology. 2001;202(2):162-6. doi: 10.1159/000051626. PMID 11306848